CLINICAL TRIAL: NCT02343679
Title: A Phase II Study of the ALK Inhibitor, Ceritinib (LDK378), in Relapsed/Refractory ALK+ Hematologic Malignancies
Brief Title: Novartis PhII Ceritinib (LDK378) in R/R ALK+ Hem Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual due to rarity of disease.
Sponsor: Anne Beaven, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Anne Beaven, MD, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056623
Record Dates: First submitted 2014-12-03; First posted 2015-01-22 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceritinib for ALK + patients (Experimental): all ALK + hematologic malignancies patients will receive ceritinib
  Interventions: Drug: ceritinib

INTERVENTIONS:
Drug: ceritinib — Ceritinib will be administered to ALK + hematologic malignancies orally at the 750mg/day dose that has been calculated as the maximum tolerated dose in prior phase I trials in lung cancer patients. Intra patient dose reductions will be allowed for toxicities. Subjects with stable disease or better will be allowed to continue study drug until disease progression or until intolerable adverse events or patient or physician choice.
  Other Names: LDK378

SUMMARY:
This is a phase II, single arm, unblinded study of ceritinib in patients with rel/ref hematologic malignancies. Up to 24 evaluable subjects will be enrolled with an interim analysis for efficacy after the first 9 subjects are enrolled. Any subject who takes at least one dose of study drug will be evaluable for safety. Only subjects who complete at least 1 cycle of study drug and have clear progression on physical exam or have had at least one restaging study will be considered evaluable for response. Each subject will receive the same dose of 750mg po daily at the study entry. Subjects with stable disease or better will be allowed to continue study drug until disease progression or until intolerable adverse events or patient or physician decision. Intrapatient dose reductions will be allowed for adverse events. This is a multicenter study with Duke as the lead site. Blood and tissue samples, will be collected and used for exploratory analysis.

DETAILED DESCRIPTION:
This is a phase II, single arm, unblinded study of ceritinib in patients with rel/ref hematologic malignancies. Up to 24 evaluable subjects will be enrolled with an interim analysis for efficacy after the first 9 subjects are enrolled. Any subject who takes at least on dose of study drug will be evaluable for safety. Only subjects who complete at least 1 cycle of study drug and have clear progression on physical exam or have had at least one restaging study will be considered evaluable for response. Each subject will receive the same dose of 750mg po daily at the study entry. Subjects with stable disease or better will be allowed to continue study drug until disease progression or until intolerable adverse events or patient or physician decision. Intrapatient dose reductions will be allowed for adverse events. Blood and tissue samples, will be collected and used for exploratory analysis.

Dose Level 0 (starting dose) 750mg/day Dose level -1 600mg/day Dose level -2 450mg/day

Baseline evaluations are to be conducted within 30 days prior to start of protocol therapy unless otherwise noted in the time to events table. Scans and x-rays must be performed within six weeks prior to the start of therapy. Bone marrow biopsy must be performed within twelve weeks prior to starting therapy. In the event that the patient's condition is deteriorating, laboratory evaluations should be repeated within 48 hours prior to initiation of the next cycle of therapy. All the labs have to be within the study eligibility range prior to the start of study treatment.

All visits should occur within 3 days before or after the scheduled day of the visit. An early or late visit will not shorten or extend the duration of that cycle - all cycles will be 28 days.

If study drug is held for any reason then the missed days should still be counted as a day in the cycle. However, if the study drug is on hold when a 28 day cycle ends, then day 1 of the next cycle and the necessary evaluations should not be started until drug is restarted. Therefore, the cycle during which a drug is held could potentially have more than 28 days.

Patients will be followed for up to 2 years after completion of therapy or until progression of disease or death, whichever comes first. In follow up, patients will be seen every 3 months for physical exam, lab draws for the first two years after completing all study drugs or until alternative therapy is begun or until progression of disease or death-whichever comes first. Radiographic imaging will be performed every 6 months for the first two years after study drug is completed.

Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event and will continue to be followed until progression of disease or death. Unacceptable adverse events are those that lead to stopping of a study drug and for which there is no resolution of drug related toxicity after a 6 week washout period so that the subject is removed from study as defined in section 6.

Patients removed from the study due to progressive disease will be followed until resolution or stabilization of any adverse events due to the agents, after which their follow up will be completed.

At a minimum, all patients who discontinue ceritinib treatment, including those who refuse to return for a final visit, will be contacted for safety evaluations during the 30 days following the last dose of treatment

ELIGIBILITY:
Inclusion Criteria:

* Alk+R/R hematologic malignancy including but not limited to ALK+ALCL or ALK+LBCL > 1 prior standard cytotoxic regimen
* Age >18
* ECOG performance status <2
* Evidence of measurable or evaluable disease
* Toxicities ≤ grade 2 due to prior therapies Exception: any grade alopecia
* Platelets >75 x 109/L
* ANC>1.5 x 109/L
* AST/ALT<3.0 x ULN, except liver involvement by their lymphoma, include if AST/ALT<5 x ULN.
* Total Bilirubin<1.5 x ULN, (includes gilbert's syndrome if total bilirubin <3.0 x ULN and direct bilirubin <1.5 x ULN)
* Potassium, magnesium, total calcium and phosphorous > lower limits of normal
* Calculated or measured CrCl> 30ml/min
* Ability to provide written informed consent
* Willing/able to comply with scheduled visits, treatment plans, laboratory tests and other procedures
* Women/men of reproductive potential must agree to use effective birth control during study and for 3 months after receiving study drug.
* Must have existing tissue available for correlative studies

Exclusion Criteria:

* No chemotherapy, radiation or surgical resection of malignancy < 3 weeks before start of study drug
* Prior therapy with other ALK inhibitor investigational agents except crizotinib
* Active, uncontrolled, serious infection or medical or psychiatric illness likely to interfere with trial
* Known HIV infection
* Extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, (history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis or clinically significant radiation pneumonitis) i.e. affecting daily living or requiring ongoing therapeutic intervention.
* Symptomatic CNS metastases and neurologically unstable or increasing doses of steroids < 2 weeks prior to study entry
* Major surgery 4 weeks before initiating protocol therapy.
* Hypersensitivity to microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide, magnesium stearate
* Diagnosis or treatment for malignancy other than NHL < 3 years before Day 1 of protocol therapy. Exceptions:

  * Basal or squamous cell carcinoma of the skin
  * In situ malignancy - completely resected.
  * Prostate cancer treated with prostatectomy or radiotherapy > 2 years before Day 1 of protocol therapy and PSA is undetectable
  * In situ malignancy - completely resected
* Current treatment with another investigational agent < 14 days before enrollment. Other non-treatment studies allowed if it won't interfere with study participation.
* Myocardial infarction or unstable angina 6 months before enrollment or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

  o QTcF>450msec
* Oral steroids > 4mg dexamethasone or equivalent/day excluding steroids used for adrenal insufficiency
* Impaired GI function from significant small bowel resection or gastric bypass surgery or inability to swallow up to five ceritinib capsules daily
* Ongoing GI adverse events > grade 2 (e.g. nausea, vomiting, or diarrhea) at start of study.
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to start of treatment and for the duration of participation:

  * Medication with a significant known risk of prolonging the QT interval or inducing Torsades de Pointes http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm
  * Strong inhibitors or strong inducers of CYP3A4/5 http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org
  * Therapeutic doses of warfarin sodium (Coumadin) or coumadin-derived anti-coagulant.
  * Enzyme-inducing anticonvulsive agents
  * Herbal supplements
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 5 years
  ORR defined as CR + PR. Stable disease of at least 3 months will also be reported.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 5 years
  Calculate the median time until disease progression or death in patients treated with ceritinib

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beaven, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States